CLINICAL TRIAL: NCT04187131
Title: An Augmented Reality Based System for Neglect Detection, Assessment, and Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Northeastern University (Other); NSF (Unknown)
Responsible Party: Principal Investigator, Murat Akcakaya, Assistant Professor, Electrical and Computer Engineering, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19060390; 1915083 (Other Grant/Funding Number: NSF)
Record Dates: First submitted 2019-12-02; First posted 2019-12-05 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- augmented reality (Experimental)
  Interventions: Behavioral: augmented reality

INTERVENTIONS:
Behavioral: augmented reality — The participants will be wearing an EEG cap and Augmented Reality headset (AR-based EEG-guided system) for 10 sessions with a licensed occupational therapist, provided in addition to usual rehabilitation care (either in inpatient rehabilitation or at home). These sessions will focus on activities of daily living that the participants want to practice. All sessions will last approximately 1 hour. These sessions will be scheduled around the existing therapy schedule to cause the least amount of interference with planned clinical activities.

SUMMARY:
The aim of this phase is to examine the feasibility and acceptability of the Augmented Reality (AR)-based and electroencephalography (EEG)-based neglect detection and rehabilitation tool.

ELIGIBILITY:
Inclusion Criteria:

* ages18 and older
* acute stroke
* admitted to inpatient rehabilitation
* presence of neglect (Behavioral Inattention Test total score <129, or scoring below pre-defined cutoff score in at least one of the six subtests)
* more than 10/% missed targets on the Augmented Reality Screening Test
* intact vibration (positive test on Vibration Sensation Test)
* intact auditory function (positive test on Auditory Sensation Test)
* English speaking

Exclusion Criteria:

* inability to follow one-step directions at least 80% of the time
* current diagnosis of dementia, Parkinson's disease, multiple sclerosis, or space-occupying tumor
* metal in the head that causes interference with the EEG system
* self-report of previous positive photic stimulation test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy; indicated by percent agreement between participant report and EEG-based assessment of neglect | week 4
  number of sessions attaining greater than 70 percentage agreement between targets identified by the participant and targets identified by EEG; participants view an augmented reality screen with randomly appearing targets in the field of view; when a target is viewed, the participant presses a keyboard key; immediately after, targets randomly appear on the augmented reality screen while the participant's brain activity is recorded by EEG; EEG detects viewed and neglected targets based on brain signals;
Reliability; indicated by correlation coefficient between two consecutive sessions of EEG recording | week 4
  number of consecutive sessions attaining Pearson correlation coefficient r greater than.10

SECONDARY OUTCOMES:
Technology Satisfaction; indicated by a mean score of 3 or higher on the Quebec User Evaluation of Satisfaction with Assistive Technology | week 4
  number of participants attaining greater than or equal to 90 percentage satisfaction; satisfaction is rated on 12 items with a 5-point likert scale, 5 indicating very high satisfaction; items are summed with total a total score of 60 indicating very high satisfaction;
Program Satisfaction; indicated by mean score of 3 or greater on the Client Satisfaction Questionnaire | week 4
  number of participants attaining greater than or equal to 90 percentage satisfaction; satisfaction is rated on 8 items with a 4-point likert scale, 4 indicating very high satisfaction; items are summed with total a total score of 32 indicating very high satisfaction;

CONTACTS AND LOCATIONS:
Overall Officials: Murat Akcakaya, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Northeastern University, Boston, Massachusetts
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Recorded EEG data may be disseminated to collaborators, other researchers, or the general public, for instance via DScholarship@Pitt: University of Pittsburgh Institutional Repository or through Pitt Box. At this time, there are no specific external parties. If in the future, access to data is requested, any identifying data to will be removed from the EEG data to protect participants' privacy.
Supporting Information: Study Protocol